CLINICAL TRIAL: NCT04926636
Title: A System and Process to Improve the Satisfaction With Hearing Health Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00010555
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Mobile App (No Intervention): This group will be supplied with Novidan DTC hearing aids and documentation following standard of care as a control. They will be provided with the mobile application allowing for the monitoring of data for study analysis and personal control of their hearing aids, but not Health and Wellness Coaching features.
- Enhanced Mobile App with Health Coaching (Experimental): This group will also be supplied with the Novidan DTC hearings aids and documentation, same as the control group, but will be supplied the enhanced mobile application that allows for participation in health coaching features. They will be assigned to a health coach and will have coaching sessions scheduled.
  Interventions: Behavioral: Health and Wellness Coaching

INTERVENTIONS:
Behavioral: Health and Wellness Coaching — An enhanced mobile application that allows for participation in health coaching features. Participants will be assigned to a health coach and will have coaching sessions scheduled.
  Arms: Enhanced Mobile App with Health Coaching

SUMMARY:
Innovative Design Labs Inc. (IDL) and its collaborators, proposes to create a cloud-based system which integrates advances and techniques from Health and Wellness Coaching (HWC) into the Hearing Aid (HA) fitting and trial process.

DETAILED DESCRIPTION:
As of 2015, 28.8 million U.S. adults could benefit from using hearing aids and the prevalence of hearing loss in the United States is predicted to rise significantly due to an aging population and the growing use of personal listening devices. However, only 28.5% of individuals who could benefit from a HA actually wears one. The non-use of hearing aids by people with hearing loss has many far-reaching implications for their physical health, mental health, and their social life. As the market moves towards a, direct-to-consumer distribution model following the 2017 FDA directive, more patients will be receiving therapy for hearing loss. While in traditional practice, an audiologist assists the patient with support adjusting to their new therapy, there is no person fulfilling that role in the direct-to-consumer model. Hypothesis: The investigators hypothesize that the integration of Health and Wellness Coaching, aided by cloud-based tools, into this process will increase patients' satisfaction and usage of hearing health products. Specific Aims: 1) Create patient/coach interaction protocol and training; 2) Develop a cloud-based Health Coaching Interface; 3) Evaluate system effectiveness through a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Significantly reduced cognitive ability (assessed using the Montreal Cognitive Assessment MoCA)
* Lack of proficiency communicating in English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
COSI Goal Achievement | 3 months
  The Client Oriented Scale of Improvement (COSI) questionnaire tracks the goals and needs of the patient through their hearing aid fitting process. Items allow the patient to qualify their degree of change for each of their needs/goals as 1) Much Worse 2) Worse 3) No Difference 4) Better 5) Much Better. Total scores are an average of item scores and range from 1 to 5 with higher scores indicating more improvement.
AQoL-8D Score | 3 months
  The Assessment of Quality of Life (AQoL) is a measure of health-related Quality of Life. AQoL-8D covers dimensions of Independent Living, Happiness, Mental Health, Coping, Relationships, Self-Worth, Pain, and Senses. Items are scored from 0 to 3. Scores range from 0 to 45 with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
Hours of Hearing Aid Use | 3 months
  Hearing aid usage information for both groups will be automatically logged on non-volatile memory inside of the hearing aid. It will record the amount of time in hours the user spent wearing their hearing aids. It is accessed and downloaded through the provided companion smartphone application.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided